CLINICAL TRIAL: NCT05475444
Title: Modified Surface of PLGA Nanoparticles in Smart Hydrogel: A Randomized Clinical Trial to Establish an Advanced Strategy Against Antibiotic Resistant Infections in Endodontics
Brief Title: PLGA Nanoparticles Entrapping Ciprofloxacin to Treat E-Fecalis Infections in Endodontics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Mona Gamal Mohamed Afifi Arafa, Associate Professor, British University In Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1643
Record Dates: First submitted 2021-02-06; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Bacterial Infections Oral

STUDY DESIGN:
Intervention Model Description: * Group I (negative control group): Root canals were not treated after cleaning and shaping.
  * Group II (positive control group): Root canals were treated with calcium hydroxide paste
  * Group III: Root canals were treated with CIP paste conventionally used by the dentist which was formed by mixing CIP with saline to form a paste.
  * Group IV: Root canals were treated with (F1) which is the prepared in-situ gel formulation containing CIP loaded chitosan coated PLGA nanoparticles.
  * Group V: Root canals were treated with (F2) which is the prepared in-situ gel containing ciprofloxacin hydrochloride.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paste and solution of ciprofloxacin as Conventional Treatment (Experimental): Paste and solution of ciprofloxacin as conventional dosage forms and drugs used to treat endodontics infections. For ciprofloxacin solution is used once daily while the paste form used weekly.
  Interventions: Device: Ciprofloxacin paste and solution
- Chitosan coated PLGA nanoparticles entrapping ciprofloxacin and incorporated in smart poloxamer gel (Experimental): Chitosan coated PLGA nanoparticles entrapping ciprofloxacin and incorporated in smart poloxamer gel dosage forms treat endodontics infections
  Interventions: Device: Chitosan Coated PLGA nanoparticles entrapping Ciprofloxacin incorporated in smart gels

INTERVENTIONS:
Device: Chitosan Coated PLGA nanoparticles entrapping Ciprofloxacin incorporated in smart gels — antibacterial nanoparticles were used because of their small size, sustained release and positive charge which interact with the negatively charged surface of bacterial cell causing its destruction.
  Other Names: Chitosan Coated PLGA nanoparticles; PLGA nanoparticles as smart gels
  Arms: Chitosan coated PLGA nanoparticles entrapping ciprofloxacin and incorporated in smart poloxamer gel
Device: Ciprofloxacin paste and solution — Conventional antibacterial paste and solution were compared to nanoparticles smart gels to treat endodontics bacterial infection
  Arms: Paste and solution of ciprofloxacin as Conventional Treatment

SUMMARY:
PLGA nanoparticles coated with Chitosan polymer were prepared and then incorporated in In -situ gel to be injected to root canals of patients suffered from bacterial infection of their endodontics.

DETAILED DESCRIPTION:
The Clinical procedures:

1. First visit Treatment plan was discussed with the patients and their acceptance to participate in the study was obtained through an informed consent.

   Coronal restorations and any carious decay were removed, teeth properly restored then rubber dam was applied for isolation. An access cavity was prepared using an appropriate size bur (Bur #3, Veterinary dental equipment, UK) , and the tooth surface was disinfected before entering the root canals using 2.5% sodium hypochlorite, then its effect was inhibited using 5% sodium thiosulphate. The old gutta percha was removed from the coronal two thirds of the root canal using bur #3 without using any solvent. Sterile saline was used for irrigation. Patency was obtained using manual k files #15 (and #10, tooth length was determined using an electronic apex locator (Electronic apex locator J Morita Root ZX, Morita Corporation, Japan). The remaining gutta percha was removed using gradually increasing sizes of manual k files (K- files, Mani, Japan) . Scrubbing of the walls using manual files was done to soak the irrigant (sterile saline) with parts of the bacterial film on the canal walls. Sterile paper point equivalent to the size of largest file reaching the working length was placed for one minute in the canal and located one millimeter away from the tooth length, this represented the first sample for bacteriological assessment (S1) then paper point was placed in 1ml sterile medium. Complete cleaning and shaping of the canal was done using 15 ml of 2.5% sodium hypchlorite as an irrigant with a side vented needle of gauge 27, placed one millimeter from the working length and manual k type files, the master apical file was determined according to each case, where its size was increased 3 times more than the initial file with obtained white dentine chips as well. After complete cleaning and shaping, the action of sodium hypochlorite was inhibited by using 10 ml of 5% sodium thiosulphate. Sodium thiosulphate was flushed from the canal using 5 ml sterile saline. A sterile paper point equivalent to the size of master apical file was placed for one minute in the canal, one millimeter away from the working length to soak the fluid and this represented the second sample for bacteriological assessment (S2), afterwards, paper point is placed in 1ml sterile medium, then the patients were randomly allocated according to the use of an intracanal medications to the five groups for 7 days. Finally, a cotton pellet and temporary filling (Orafill-G) was applied under complete aseptic conditions
2. Second visit

   • Assessment of the clinical signs and symptoms was done.
3. Clinical criteria for healing:

1. No pain with percussion 2. No pain with palpation 3. Tooth asymptomatic and functional If the patient showed these clinical findings, root canals were obturated. If the patient had all or one of them, cleaning, shaping and medication steps were repeated and the patient re-scheduled for another visit after 7 days. If the patient was asymptomatic and the tooth was functional, then a temporary filling was removed under rubber dam isolation. Twenty ml of sterile saline was used to remove the intracanal medicaments until it got out clear from the canal then sterile paper point was placed in the canal one millimeter away from the working length to take the last sample (S3), paper point was placed in 1ml sterile medium, finally master cone adjustment and obturation were done.

These sterile paper points with three samples (S1, S2, S3) were placed separately in sterile falcon tubes, labeled according to the type of medication and the order of the sample. One ml of sterile tryptic soy broth (TSB) supplemented with 0.5% glucose (TSBG) was added to each tube , then tubes were transferred to the microbiology lab within 2-3 hours from sampling procedure in an ice box 4.Microbiological evaluation All microbiological steps were performed in the vicinity of a trilaminar flow cabinet to avoid air contamination of the samples.

5. Total percentage of bacterial reduction: A total of 100 μl from each sample containing (4mg) drug in addition to Ca (OH)2 paste and (4mg) CIP past were aspirated using a sterile micropipette from each tube. A sterile inoculum was used to add samples to the brain heart media. The samples were labeled according to the groups of medication and incubated for 24 hours at 37 ºC. After incubation, the total number of bacterial counts was estimated

ELIGIBILITY:
Inclusion Criteria:

* Root canal filled single rooted teeth with post treatment disease manifested by one or more of the following signs and symptoms:
* History of recurrent acute and/or chronic periapical abscess
* Pain on palpation and/or percussion at least after one month of previous procedure
* Radiographic evidence of bone loss either as a new developing lesion or an increase in the size of a pre-existing one.

Exclusion Criteria:

* Teeth that were badly broken down indicated for extraction or with difficult isolation
* Immuno-compromised patients.
* Patients with history of taking antibiotics orally.
* Periodontally affected teeth.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Determination of Bacterial count by counting bacterial colonies of the sample | One week
  Bacterial count was expected to be decreased by counting bacterial colonies of the sample after treatment and comparing with control without treatment

SECONDARY OUTCOMES:
Determination of the Biofilm inhibition using crystal violet and microplate reader | one week
  Biofilm is to be inhibited and being small by using of stains crystal violet as marker, in order to more accurately identify cells of interest and distinguish from culture debris.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Arafa, Professor, Principal Investigator — The British University in Egypt
Locations (1):
- Mona Arafa, Cairo, El Sherouk City , Suez Desert Road , Cairo - P.O. Box 43, Egypt

IPD SHARING:
Plan to Share IPD: No